CLINICAL TRIAL: NCT06272435
Title: Beverage Hydration Index: Assessment of Four Rehydration Solutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2024-64
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hydration
Keywords: Liquid IV; Electrolyte; Beverage Hydration Index
MeSH Terms: interventions — Amino Acids; Water

STUDY DESIGN:
Intervention Model Description: Semi-blinded, placebo controlled, crossover design
Who Masked: Participant
Masking Description: Treatments will be labeled A-D. Subjects will be provided prepared beverages prepared in cup.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (24):
- Water, Multiplier, Sugar with Amino Acids, and Sugar Free (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Water, Multiplier, Sugar Free, and Sugar with Amino Acids (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Water, Sugar with Amino Acids, Multiplier, and Sugar Free (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Water, Sugar with Amino Acids, Sugar Free, and Multiplier (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Water, Sugar Free, Multiplier, and Sugar with Amino Acids (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Water, Sugar Free, Sugar with Amino Acids, and Multiplier (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Multiplier, Water, Sugar with Amino Acids, and Sugar Free (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Multiplier, Water, Sugar Free, and Sugar with Amino Acids (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Multiplier, Sugar with Amino Acids, Water, and Sugar Free (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Multiplier, Sugar with Amino Acids, Sugar Free, and Water (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Multiplier, Sugar Free, Water, and Sugar with Amino Acids (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Multiplier, Sugar Free, Sugar with Amino Acids, and Water (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar with Amino Acids, Water, Multiplier, and Sugar Free (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar with Amino Acids, Water, Sugar Free, and Multiplier (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar with Amino Acids, Multiplier, Water, and Sugar Free (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar with Amino Acids, Multiplier, Sugar Free, and Water (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar with Amino Acids, Sugar Free, Water, and Multiplier (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar with Amino Acids, Sugar Free, Multiplier, and Water (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar Free, Water, Multiplier, and Sugar with Amino Acids (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar Free, Water, Sugar with Amino Acids, and Multiplier (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar Free, Multiplier, Water, and Sugar with Amino Acids (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar Free, Multiplier, Sugar with Amino Acids, and Water (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar Free, Sugar with Amino Acids, Water, and Multiplier (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water
- Sugar Free, Sugar with Amino Acids, Multiplier, and Water (Experimental): Subjects will follow control diet for 24 hours prior to visit. At the study visit, baseline measures will be collected prior to treatment. Subjects will then consume the assigned treatment (one treatment per visit in order above) and additional experimental measurements will be collected.
  Interventions: Dietary Supplement: Multiplier; Dietary Supplement: Sugar Free; Dietary Supplement: Sugar Free with Amino Acids; Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Multiplier — Subjects will consume 1 Liter (2 servings) of commercially available Hydration Multiplier product at a rate of 250 milliliters per 7.5 minutes.
Dietary Supplement: Sugar Free — Subjects will consume 1 Liter (2 servings) of experimental Sugar Free Hydration Multiplier product at a rate of 250 milliliters per 7.5 minutes.
Dietary Supplement: Sugar Free with Amino Acids — Subjects will consume 1 Liter (2 servings) of commercially available Sugar Free Hydration Multiplier product that contains amino acids at a rate of 250 milliliters per 7.5 minutes.
Dietary Supplement: Water — Subjects will consume 1 Liter of water at a rate of 250 milliliters per 7.5 minutes.

SUMMARY:
No studies to date to evaluate the effects of the three different liquid IV electrolyte products on the beverage hydration index (BHI). Therefore, the purpose of this study is to determine the impact of three different LIV products (Hydration multiplier, Sugar Free formulation with Amino Acids, and Sugar Free with allulose) on hydration status in young and active men and women compared to a control (water). The study will follow the same approach as used by Maughan and colleagues (2016) to measure the fluid balance (the difference between the amount of water consumed and passed as urine) and BHI (the relative amount of urine passed after consumption of a drink compared to water) including time in positive fluid balance, as well as determining electrolyte concentrations, osmolality, specific gravity, and sodium and potassium in urine.

DETAILED DESCRIPTION:
Many attempts have been made to improve and measure the hydration status of active individuals. This typically involves the ingestion of fluids leading up to activity (typically plain water), as well as the ingestion of fluids during the activity itself (water, along with a diluted carbohydrate/electrolyte beverage). This approach seems to work well; however, some debate remains over what the best fluid is to consume, in particular related to the macronutrient type and the specific electrolyte mix.

No studies to date to evaluate the effects of the three different liquid IV electrolyte products on the beverage hydration index (BHI). Therefore, the purpose of this study is to determine the impact of three different LIV products (Hydration multiplier, Sugar Free formulation with Amino Acids, and Sugar Free with allulose) on hydration status in young and active men and women compared to a control (water). The study will follow the same approach as used by Maughan and colleagues (2016) to measure the fluid balance (the difference between the amount of water consumed and passed as urine) and BHI (the relative amount of urine passed after consumption of a drink compared to water) including time in positive fluid balance, as well as determining electrolyte concentrations, osmolality, specific gravity, and sodium and potassium in urine.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) <35 kilgrams per square meter
* consistent dietary intake and exercise throughout study period
* consumes 2 liters (women) or 2.5 liters (men) of water per day prior to study visits
* able to fast for 15 hours

Exclusion Criteria:

* sensitivity or be allergic to any components of the study product they will be excluded.
* tobacco user
* specialized diet (low carbohydrate/ketogenic diet, carnivore diet, intermittent fasting, etc.)
* caffeine consumption within 12 hours of study visit
* strenuous activity within 24 hours of study visit
* history or presence of a clinically relevant (that required or requires treatment) cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder
* conditions that alter fluid balance or electrolytes/hydration status
* consuming any medication which may alter fluid retention/electrolyte levels such as sodium-glucose co-transporter 2 (SGLT2) inhibitor (for type 2 diabetes), laxatives, diuretics, Apremilast, chemotherapy, or lithium.
* consuming nutritional supplements, performance enhancing drugs, and/or non-steroidal anti-inflammatory drugs within 7 days of study visits excluding screening).
* employee of Liquid IV
* be enrolled in another clinical study within 30 days of the first study visit
* active infection or illness of any kind

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Beverage Hydration Index | 0 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage Hydration Index | 60 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage Hydration Index | 120 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage Hydration Index | 180 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.
Beverage Hydration Index | 240 minutes after beverage consumption
  Beverage Hydration index calculated as mass of urine collected following control (water) consumption divided by the mass of urine collected following treatment.

SECONDARY OUTCOMES:
Net Fluid Balance | 0 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 60 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 120 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 180 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Net Fluid Balance | 240 minutes after beverage consumption
  Net Fluid balance will be calculated subtracting total urine collected from total liquid consumed
Urine Osmolality | 0 minutes before beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 0 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 60 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 120 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 180 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Osmolality | 240 minutes after beverage consumption
  Urine Osmolality will be measured in milliosmoles per kilogram of water.
Urine Sodium | 0 minutes before beverage consumption
  Urine Sodium will be measured in millimoles per liter.
Urine Sodium | 0 minutes after beverage consumption
  Urine Sodium will be measured in millimoles per liter.
Urine Sodium | 60 minutes after beverage consumption
  Urine Sodium will be measured in millimoles per liter.
Urine Sodium | 120 minutes after beverage consumption
  Urine Sodium will be measured in millimoles per liter.
Urine Sodium | 180 minutes after beverage consumption
  Urine Sodium will be measured in millimoles per liter.
Urine Sodium | 240 minutes after beverage consumption
  Urine Sodium will be measured in millimoles per liter.
Urine Potassium | 0 minutes before beverage consumption
  Urine Potassium will be measured in millimoles per liter.
Urine Potassium | 0 minutes after beverage consumption
  Urine Potassium will be measured in millimoles per liter.
Urine Potassium | 60 minutes after beverage consumption
  Urine Potassium will be measured in millimoles per liter.
Urine Potassium | 120 minutes after beverage consumption
  Urine Potassium will be measured in millimoles per liter.
Urine Potassium | 180 minutes after beverage consumption
  Urine Potassium will be measured in millimoles per liter.
Urine Potassium | 240 minutes after beverage consumption
  Urine Potassium will be measured in millimoles per liter.
Urine Specific Gravity | 150 minutes before beverage consumption
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 0 minutes before beverage consumption urine
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 0 minutes after beverage consumption urine
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 60 minutes after beverage consumption urine
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 120 minutes after beverage consumption urine
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 180 minutes after beverage consumption urine
  Urine Specific Gravity will be measured via refractometry.
Urine Specific Gravity | 240 minutes after beverage consumption urine
  Urine Specific Gravity will be measured via refractometry.
Sodium balance | 0 minutes after beverage consumption
  Sodium Balance will be calculated subtracting total sodium in urine from total sodium consumed in beverage.
Sodium balance | 60 minutes after beverage consumption
  Sodium Balance will be calculated subtracting total sodium in urine from total sodium consumed in beverage.
Sodium balance | 120 minutes after beverage consumption
  Sodium Balance will be calculated subtracting total sodium in urine from total sodium consumed in beverage.
Sodium balance | 180 minutes after beverage consumption
  Sodium Balance will be calculated subtracting total sodium in urine from total sodium consumed in beverage.
Sodium balance | 240 minutes after beverage consumption
  Sodium Balance will be calculated subtracting total sodium in urine from total sodium consumed in beverage.
Potassium balance | 0 minutes after beverage consumption
  Potassium Balance will be calculated subtracting total potassium in urine from total potassium consumed in beverage.
Potassium balance | 60 minutes after beverage consumption
  Potassium Balance will be calculated subtracting total potassium in urine from total potassium consumed in beverage.
Potassium balance | 120 minutes after beverage consumption
  Potassium Balance will be calculated subtracting total potassium in urine from total potassium consumed in beverage.
Potassium balance | 180 minutes after beverage consumption
  Potassium Balance will be calculated subtracting total potassium in urine from total potassium consumed in beverage.
Potassium balance | 240 minutes after beverage consumption
  Potassium Balance will be calculated subtracting total potassium in urine from total potassium consumed in beverage.
Body Mass | 0 minutes before beverage consumption
  Body Mass in kilograms will be measured using a digital scale
Body Mass | 240 minutes after beverage consumption
  Body Mass in kilograms will be measured using a digital scale
Mood and Digestive Questionnaire | 0 minutes before beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 0 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 60 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 120 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 180 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)
Mood and Digestive Questionnaire | 240 minutes after beverage consumption
  Subjects will be asked to self-assess their mood and digestive state via a visual analog scale questionnaire with scale 0 (None) to 10 (Extreme)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — Center for Nutraceutical and Dietary Supplement Research
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No